CLINICAL TRIAL: NCT03602391
Title: The Senior Companion Program Plus (SCP Plus): A Psychoeducational Intervention for African American Dementia Caregivers
Brief Title: The Senior Companion Program Plus
Acronym: SCP Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Noelle Fields, Assistant Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0431
Record Dates: First submitted 2018-07-06; First posted 2018-07-26 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Family; Alzheimer Dementia
MeSH Terms: conditions — Alzheimer Disease | interventions — Urocortins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCP Plus (Experimental)
  Interventions: Behavioral: SCP Plus
- Services as usual (No Intervention)

INTERVENTIONS:
Behavioral: SCP Plus — The primary goal of the proposed project is to develop an in-home psychoeducational intervention (Senior Companion Program Plus, or SCP Plus) that is accessible, affordable, and sustainable for low-income African American ADRD caregivers. A weekly, 60 minute psychoeducational module will be delivered face-to-face across 9 weeks and will focus on education about ADRD, behavior management, communication skills, and aspects of providing care that enhance meaning such as spirituality. In order to provide an accessible intervention that is potentially sustainable, Senior Companions will be trained to provide the intervention in the homes of the African American ADRD caregivers.
  Arms: SCP Plus

SUMMARY:
Alzheimer's disease and related dementia (ADRD) is one of the most challenging chronic health conditions in the United States and considerable disparities exist in the diagnosis and prevalence of ADRD among communities of color. Research suggests that ADRD caregiver interventions have demonstrated efficacy, however, it remains unknown whether existing ADRD caregiver interventions are useful or accessible to African American ADRD caregivers in community settings.

The primary goal of the proposed project is to develop an in-home psychoeducational intervention (The Senior Companion Program Plus, or SCP Plus) that is accessible, sustainable, and affordable for African American ADRD caregivers. The SCP Plus will focus on African American ADRD caregivers who are particularly affected by poverty, discrimination, and barriers to health care services and supports. A recent pilot study has established the feasibility and utility of SCP Plus. With the assistance of 6 student research assistants over the course of the project, we will implement the SCP Plus at sites in Texas, Louisiana, and Arkansas, recruiting approximately 114 participants. The participants will be randomized with 57 caregivers receiving the SCP Plus and 57 caregivers receiving services as usual with the Senior Companion Program. A weekly, 60 minute psychoeducational module will be delivered face-to-face across 9 weeks and will focus on education about ADRD, behavior management, communication skills, and aspects of providing care that enhance meaning such as spirituality. In order to provide an accessible and cost effective intervention that is potentially sustainable, senior companions will be trained to provide the intervention in the homes of the African American ADRD caregivers.

Specific Aim 1. Determine whether SCP Plus reduces level of burden and stress among African American caregivers over a 3- and 6-month period when compared to a usual care control group.

Specific Aim 2. Ascertain if SCP Plus improves coping skills among African American caregivers over a 3- and 6-month period when compared to a usual care control group.

Specific Aim 3. Examine whether SCP Plus improves the level of satisfaction with support social among African American caregivers over a 3- and 6- month period when compared to a usual care control group.

Specific Aim 4. Explore and interpret the statistical results obtained in the first quantitative phase to help explain why participants who scored in the lower and upper quartiles on caregiver burden/stress were impacted or not by the usefulness of the intervention.

Successful design, delivery, and evaluation of the SCP Plus will lead to a cost effective, sustainable, and accessible intervention that can be implemented in other Senior Companion programs across the country, thus maximizing its impact as a community-based program to address the needs of African American ADRD caregivers.

ELIGIBILITY:
Inclusion Criteria:

A. Senior Companions have to be currently participating in the Senior Companions Program B. Senior Companions have to be currently providing respite services to the caregivers C. Family caregivers must self-identify as African American D. Family caregivers must be at least 21 years of age E. Family caregivers must provide unpaid care for an older adult with ADRD F. The persons with ADRD must have a physician diagnosis of ADRD and live at home in the community.

G. The capacity for and willingness to provide written informed consent, to accept the randomized group assignment, to attend all study related visits, and to comply with the study protocol.

Exclusion Criteria:

A. Family caregivers who are involved in another caregiver psychosocial intervention study or have an acute illness that would prevent them from participating for at least 6 months will not be eligible.

B. Self-identified non-African American caregivers will be excluded from enrollment in the study, because of the specificity of the cultural components of the Senior Companion Program Plus being tested.

C. Senior Companions who are not serving a client with ADRD from African American backgrounds will be excluded as the Senior Companion Program Plus is designed for dementia family caregivers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Senior Source, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fields NL, Xu L, Williams IC, Gaugler JE, Cipher DJ. The Senior Companion Program Plus for African American Caregivers of Persons With Alzheimer Disease and Related Dementias: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Jul 24;12:e49679. doi: 10.2196/49679. PMID 37486759

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The original participant enrollment goal was 114 participants. However, due to COVID-19, only 20 participants consented and were enrolled in the study.
Groups:
- SCP Plus Intervention: SCP Plus: The primary goal of the proposed project is to develop an in-home psychoeducational intervention (Senior Companion Program Plus, or SCP Plus) that is accessible, affordable, and sustainable for low-income African American ADRD caregivers. A weekly, 60 minute psychoeducational module will be delivered face-to-face to African American ADRD caregivers across 9 weeks and will focus on education about ADRD, behavior management, communication skills, and aspects of providing care that enhance meaning such as spirituality. In order to provide an accessible intervention that is potentially sustainable, Senior Companions, who are volunteers as part of the AmeriCorps Seniors Program, will be trained to provide the intervention in the homes of the African American ADRD caregivers. The care recipients (CR) with ADRD are not included as participants in the study.
- Services as Usual: This group receives services as usual from the Senior Companion Program. Services as usual means that the Senior Companion provides respite to the family caregiver. The care recipient (CR) with ADRD is not included as a participant in the study.
Period: Overall Study
Arm/Group | SCP Plus Intervention | Services as Usual
Started | 11 | 9
Completed | 4 | 3
Not Completed | 7 | 6
Not completed — COVID-19 | 7 | 6

BASELINE CHARACTERISTICS:
Population: These numbers refers to the African American ADRD caregivers in the study. The care recipients with ADRD are not part of the study as the intervention is a pschoeducational intervention for ADRD caregivers. Any mention of a dyad is the Senior Companion-caregiver. However, our outcomes are focused only on the ADRD caregiver as they are the target of the psychoeducational intervention. "Services as usual" refers to the ADRD caregivers who are receiving respite from the Senior Companion.
Groups:
- Services as Usual: Participants will receive services as usual from the Senior Companion Program.
- Total: Total of all reporting groups
Arm/Group | SCP Plus | Services as Usual | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Median (Full Range); unit: years] | 62 [48 to 71] | 58 [41 to 80] | 60.5 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 9 | 20
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20
Self-rated health [Median (Full Range); unit: units on a scale] — A single item that asks the ADRD caregiver, "In general, would you say your health is poor, fair, good, very good, or excellent?" Response for each item on the 5-point scale include: (1 = poor; 2 = fair; 3 = good; 4= very good; 5 = excellent) with higher score representing greater self-reported health. Researchers calculated a score for each ADRD caregiver by using the response to that single item and overall median of participants is reported. All survey data collection involved a researcher asking the ADRD caregiver the survey questions over the telephone and documenting their responses.
  units on a scale | 3 [1 to 4] | 3 [2 to 5] | 3 [1 to 5]
Financial strain [Median (Full Range); unit: units on a scale] — A single item that asks the ADRD caregiver, "Do you feel difficult in paying for basic needs such as food, housing, medical care, and heating? " Response for each item on the 3-point scale include: (0 = not difficult at all; 1 = a little difficult; 2 = difficult; 3 = very difficult) with higher score representing greater financial strain. Researchers calculated a score for each ADRD caregiver by using the response to that single item and overall median of participants is reported. All data collection involved a researcher asking the ADRD caregiver the survey questions over the telephone.
  units on a scale | 3 [0 to 3] | 2 [1 to 3] | 3 [0 to 3]
Marital status [Count of Participants; unit: Participants]
  Married | 5 | 6 | 11
  Divorced | 4 | 1 | 5
  Widowed/Other | 2 | 2 | 4
Living arrangement [Median (Full Range); unit: people living in household] | 2 [0 to 4] | 2 [1 to 7] | 2 [0 to 7]
Education [Count of Participants; unit: Participants]
  High school graduate or below | 6 | 2 | 8
  Some college | 4 | 6 | 10
  College graduation or above | 1 | 1 | 2
Employment [Count of Participants; unit: Participants]
  Full employment | 3 | 6 | 9
  Part-time employment | 4 | 1 | 5
  Retired/Unemployed | 4 | 2 | 6
Religiosity [Median (Full Range); unit: units on a scale] — Six items that ask the ADRD caregiver about their religious or spiritual beliefs. All items have a 4-point scale ranging from 1 (not at all), 2 (somewhat), 3 (quite a bit), and 4 (a great deal) with higher score representing greater religiosity. Median of the 6 items is analyzed. Overall median of participants is reported. All survey data collection involved a researcher asking the ADRD caregiver the survey questions over the telephone and documenting their responses.
  units on a scale | 3 [1 to 4] | 4 [3 to 4] | 3.5 [1 to 4]
Relationship to the care recipient [Count of Participants; unit: Participants]
  Spouse | 1 | 0 | 1
  Adult child | 6 | 7 | 13
  Sibling/other | 4 | 2 | 6
Length of care [Median (Full Range); unit: years] | 5 [3 to 12] | 5 [1 to 26] | 5 [1 to 26]
Use of formal services [Count of Participants; unit: Participants] — The single item question asks the ADRD caregiver: How frequently do you receive formal services (nurse, senior companions, etc.)?
  Participants
    Once or less than once a week | 0 | 1 | 1
    Several times a week | 10 | 6 | 16
    Every day | 1 | 2 | 3
Satisfaction with formal services [Count of Participants; unit: Participants]
  Unsatisfied | 1 | 1 | 2
  Satisfied | 8 | 4 | 12
  Strongly satisfied | 2 | 4 | 6
Daily care hours [Median (Full Range); unit: hours per day] | 12 [2 to 24] | 12 [3 to 24] | 12 [2 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Change in Caregiver Burden and Stress
Description: The 22-item version of the Zarit Burden Interview (ZBI) will be used to test caregiver stress and/or burden. The ZBI was developed to measure burden among caregivers of community-dwelling persons with dementia. The items are scored from 0 (never); 1 (rarely); 2 (sometimes); 3 (quite frequently); 4 (nearly always) with higher scores indicating higher levels of distress. Total scores can range from 0 to 88. Median of the 22 items is analyzed. Overall median of participants is reported. All survey data collection involved a researcher asking the ADRD caregiver the survey questions over the telephone and documenting their responses.
Time Frame: pre, post, 6-month follow up
Population: Analysis population is the same as those who were enrolled, completed a baseline survey, completed the intervention, and remained in the study for the 6 month follow-up.
Measure: Median (Full Range); unit: score on a scale
Groups:
- SCP Plus Intervention: SCP Plus: The primary goal of the proposed project is to develop an in-home psychoeducational intervention (Senior Companion Program Plus, or SCP Plus) that is accessible, affordable, and sustainable for low-income African American ADRD caregivers. A weekly, 60 minute psychoeducational module will be delivered face-to-face across 9 weeks and will focus on education about ADRD, behavior management, communication skills, and aspects of providing care that enhance meaning such as spirituality. In order to provide an accessible intervention that is potentially sustainable, Senior Companions will be trained to provide the intervention in the homes of the African American ADRD caregivers.
- Services as Usual: This group receives services as usual from the Senior Companion Program.
Arm/Group | SCP Plus Intervention | Services as Usual
Number analyzed (Participants) | 4 | 3
score on a scale
  Pre-test | 40 [16 to 63] | 18 [8 to 44]
  Post-test | 32 [10 to 45] | 18.5 [12 to 39]
  6-month follow up | 15 [13 to 30] | 7 [4 to 10]

2. Primary Outcome: Change in Caregiver Coping Skills
Description: The Brief Cope Scale will be used to measure coping skills. The Brief Cope questionnaire consists of 28 items measuring the ways/strategies caregivers have been coping with the stress in their life with 4-point scale ranging from "I have not been doing this at all"(1) to "I have been doing this a lot" (4). This Brief Cope scale consists of 14 subscales (with 2 items for each subscale). Sum scores for each subscale will be calculated, ranging from 2 to 8, with higher scores indicating better coping skills. A final total sum score will also be calculated by combining all the sum scores of the 14 subscales, ranged from 28 to 112. The higher the total scores, the better the coping skills.
Time Frame: pre, post, 6-month follow up
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | SCP Plus Intervention | Services as Usual
Number analyzed (Participants) | 4 | 3
score on a scale
  Pre-test | 81 [55 to 93] | 73 [67 to 98]
  Post-test | 96 [74 to 101] | 82 [74 to 98]
  6-month Follow up | 79 [72 to 94] | 90 [61 to 101]

3. Primary Outcome: Change in Caregiver Level of Satisfaction With Social Support
Description: Levels of satisfaction with social support was measured by asking caregivers 4 questions about how they feel satisfied with the support they received in the past month from friends, family, and others regarding: (1) overall help from friends and family, (2) help with transportation, housework and yard work, and shopping from friends and family; (3) help with support, comfort, interest and concern from others, (4) suggestions, clarifications, and sharing of similar experiences from others. Each item was measured with 3 Likert scale ranged from (0) 'Not at all', (1) 'a little', (2) 'moderately', to (3) 'very'. The sum score ranged from 0-12 with higher scores indicating higher level of satisfaction with social support. Overall median of participants is reported. All survey data collection involved a researcher asking the ADRD caregiver the survey questions over the telephone and documenting their responses.
Time Frame: pre, post, 6-month follow up
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | SCP Plus Intervention | Services as Usual
Number analyzed (Participants) | 4 | 3
score on a scale
  Pre-test | 3.5 [0 to 6] | 9 [5 to 12]
  Post-test | 4 [3 to 12] | 12 [9 to 12]
  6-month follow up | 11.5 [5 to 12] | 12 [9 to 12]

ADVERSE EVENTS:
Time Frame: 6 months
Description: No adverse events were suspected to be caused by study intervention/procedures.
Arm/Group | SCP Plus Intervention | Services as Usual
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

LIMITATIONS AND CAVEATS:
The results of this study must be interpreted with caution, as there are several limitations that provide lessons for future studies. The final sample size was very small, due in part to the negative impact of COVID-19. Due to the challenges and risks of conducting an in-person intervention during COVID-19, data collection was suspended in March 2020. Therefore, we could not control for any confounding variables when examining the preliminary effectiveness of the SCP Plus program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT03602391/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT03602391/ICF_001.pdf